CLINICAL TRIAL: NCT04229160
Title: Noninvasive 3D Mapping in Persistent Atrial Fibrillation, to Describe Modifications of the Arrhythmogenic Substrate After Pulmonary Vein Isolation and Identify Potential Predicting Factors of Ablation Success
Acronym: CRYOVEST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/0418/HP
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation, Persistent
Keywords: pulmonary vein isolation; cardioversion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with persistent atrial fibrillation (Experimental): persistent atrial fibrillation is defined as lasting longer than 6 months documented by a 24h holter monitoring
  Interventions: Device: Noninvasive mapping (Cardioinsight® system); Device: long-term cardiac monitoring (LINQ system); Procedure: Atrial Fibrillation ablation procedure

INTERVENTIONS:
Device: Noninvasive mapping (Cardioinsight® system) — Noninvasive mapping (Cardioinsight® system) of the left atria before the Atrial fibrilation ablation procedure
Device: long-term cardiac monitoring (LINQ system) — long-term cardiac monitoring (LINQ system) is used to evaluate recurrence rate following AF ablation procedure
Procedure: Atrial Fibrillation ablation procedure — Atrial Fibrillation ablation procedure is done with standard practice

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia in adults. It is a major cause of ischemic stroke and heart failure. Intravascular cardiac ablation of the left atrium by catheter delivery is an efficient treatment to restore sinus rhythm. AF ablation is a class IIa treatment for patients with symptomatic persistent AF refractory or intolerant to antiarrhythmic medication. There are still many debates considering the ablation strategy. The pulmonary veins remain the cornerstone of AF ablation therapy, even in persistent AF. There is a large electrical remodeling occurring in the left atrium between paroxysmal AF, early persistent AF and long-standing persistent AF. However, no multicentric and randomized study has demonstrated so far the interest of targeting other left atrial substrate, such as rotors or focal sources.

Our study aims to describe with a noninvasive mapping system the arrhythmogenic substrate of persistent AF > 6 months pre- and post-cardioversion, and after pulmonary vein isolation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented persistent Atrial Fibrillation lasting longer than 6 months documented by 24h holter monitoring
2. Age between 18 and 75 years
3. Efficient oral anticoagulation during at least 1 month before the procedure
4. Social security affiliation
5. Feasible patient follow-up
6. Patient willing to comply with study requirements and give informed consent to participate in this clinical study
7. Indication for Pulmonary Vein isolation

Exclusion Criteria:

1. Previous atrial fibrillation ablation
2. Previous left atrial ablation or surgery
3. Atrial fibrillation without spontaneous RR interval > 1000ms and with LVEF < 35% (measured by TTE)
4. Presence of a mechanical mitral valve
5. Current intracardiac thrombus
6. Any condition contraindicating chronic anticoagulation
7. Uncontrolled hyperthyroidism
8. Anteroposterior LA diameter > 55 mm measured by TTE
9. Body mass index ≥ 40 kg/m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-09 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2026-06-24 (Estimated)

PRIMARY OUTCOMES:
Number of focal sources and rotors in atrial segments | within 1 hour post-cardioversion procedure
Number of focal sources and rotors in atrial segments | within 1 hour post-Pulmonary Vein Isolation procedure

SECONDARY OUTCOMES:
Number of Atrial Fibrillation recurrence following AF ablation procedure | 1 year post-procedure
Number of success of Atrial Fibrillation induction after initial electrical cardioversion | within 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ANSELME, Pr, Principal Investigator — University Hospital, Rouen
Locations (4):
- France (4):
  - Caen University Hospital, Caen
  - Dieppe Hospital, Dieppe
  - Groupe Hospitalier du Havre, Le Havre
  - Rouen University Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No